CLINICAL TRIAL: NCT06038110
Title: Use of Axillary Ultrasound to Guide Breast Cancer Management in the Genomic Assay Era: A Retrospective Cohort Study
Brief Title: Use of Axillary Ultrasound to Guide Breast Cancer Management in the Genomic Assay Era
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: CIRB Ref:2022/2514
Record Dates: First submitted 2023-09-06; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Axillary Ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: axillary ultrasound — usefulness of axillary ultrasound in predicting need for chemotherapy or upfront surgery

SUMMARY:
The investigators aimed to determine if axillary ultrasound can reliably distinguish between patients with limited or high nodal burden, so that the patients with limited nodal burden can potentially avoid chemotherapy and instead receive upfront surgery followed by gene assay testing.

ELIGIBILITY:
Inclusion Criteria:

* breast cancer patients with T1-3, HR-positive and HER2-negative disease.
* aged≥ 50 years old
* had axillary ultrasound prior to operation
* axillary lymph node dissection

Exclusion Criteria:

* Patients with neoadjuvant chemotherapy
* bilateral cancers

Ages: 21 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients with T1-3, HR-positive and HER2-negative disease, aged≥ 50 years old, had axillary ultrasound prior to operation and axillary lymph node dissection
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2007-01-01 (Actual); Primary Completion 2024-01-31 (Estimated); Study Completion 2024-01-31 (Estimated)

PRIMARY OUTCOMES:
the number of abnormal nodes on ultrasound | from the date of diagnosis to the date of surgery, up to 12 weeks
  the number of abnormal nodes on ultrasound which was done at the time of diagnosis will be measured

CONTACTS AND LOCATIONS:
Locations (1):
- KK Women's and Children's Hospital, Singapore, Singapore